CLINICAL TRIAL: NCT05850013
Title: The Measurement of Vital Signs in Children by Lifelight® Software in Comparison to the Standard of Care The VISION-Junior Study
Brief Title: The Measurement of Vital Signs in Children by Lifelight® Software in Comparison to the Standard of Care
Acronym: VISION-Jr
Status: Completed | Type: Observational
Sponsor: Xim Limited (Industry)
Collaborators: South Tyneside and Sunderland NHS Foundation Trust (Other); Mind Over Matter Medtech Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: IRAS Reference: 321956
Record Dates: First submitted 2023-02-10; First posted 2023-05-09 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Cardiovascular Diseases; Respiratory Disease; Febrile Illness; Pediatric ALL
Keywords: video; audio; vital signs
MeSH Terms: conditions — Cardiovascular Diseases; Respiration Disorders; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Sub Protocol 1: Sub protocol 1 - Blood pressure measured in participants who are able to cooperate and are relatively still Within each study session, compliant participants will have their blood pressure measured using standard-of-care equipment and methods during the same 60 seconds that their other vital signs are measured
  Interventions: Device: Lifelight Junior
- Sub protocol 2: OPTIONAL Sub protocol 2: Electrocardiogram (ECG) for measurement of Heart rate variability This sub-protocol is relevant for children who would benefit from having a 3-lead ECG to capture beat to beat variability. This will be done in a subset of the participants, and ideally on a subsequent that is representative of the full cohort of participants in terms of age profile, skin tone distribution and illness.
  Interventions: Device: Lifelight Junior
- Sub protocol 3: The questionnaire will ask questions related to vital sign monitoring habits and preferences, or not, of Lifelight®-type technologies for measuring vital signs instead of standard-of-care methods.
  Interventions: Device: Lifelight Junior

INTERVENTIONS:
Device: Lifelight Junior — Lifelight® is an app developed by xim that measures VS including heart rate, respiratory rate and blood pressure. All you need to do to have these vital signs measured is look at your smartphone or tablet camera for 20-40 seconds. The app has used data from over 1 million heartbeats to learn how to measure these vital signs in adults. The technology is already available for doctors and nurses to use with adult patients in some specific scenarios

SUMMARY:
A prospective basic science study for collection of training and testing data for development of Lifelight® Junior

DETAILED DESCRIPTION:
This study will be hospital-based, including paediatric emergency department (PED), inpatient wards and outpatient departments).

The participants will have their vital signs (such as heart rate, respiratory rate, oxygen saturation, blood pressure and temperature) measured using standard-of-care methods. Concurrent with this, videos of the participants' face/torso, and audio of the sounds made by the participants (cry, wheeze, cough) will be recorded. These data will later be used to train the Lifelight® Junior algorithms so that the technology can help in detection of illness and deterioration in children.

Primary Objective Collect the data needed to develop Lifelight® Junior so that it can measure the heart rate, respiratory rate and oxygen saturation of children.

Secondary Objective

1. Assess the feasibility of developing other (direct or indirect) measurement functions in Lifelight® Junior, including temperature, blood pressure, heart rate variability and audio analysis (cry, wheeze, cough).
2. Evaluate the impact of subject-specific variables on the vital sign measurements e.g., medication, cosmetics, facial/body hair and skin tone.
3. Obtain data to understand patient and parent/guardian/carer vital sign measurement habits and preferences
4. Assess the usability of Lifelight® Junior for measuring vital signs in children

To ensure the study collects data that can train Lifelight® Junior in an efficient way, the recruitment should be divided as follows:

* At least 12% of study participants should fall into each of the following age bands:

  * Age 0-1
  * Age 1-2
  * Age 2-5
  * Age 5-11
  * Age 11-14
  * Age 14-18
* At least 40% of the study participants shall be male and at least 40% shall be female.
* At least 40% of the study participants shall be each of the following:

  * Febrile (≥ 38°C) measured how?
  * Afebrile
  * Ill (as judged by the clinical staff), of whom at most 50% shall have an acute respiratory illness e.g., bronchiolitis, asthma, viral induced wheeze, pneumonia, croup, etc.
  * Well, including children with a minor injury

Ideally, 15% of participants should have a Fitzpatrick skin tone of 4, 5 or 6 First reference to this - need to bring it in earlier and to reference it. However, this is not a hard target as achieving this figure is dependent on the demographic diversity of the study region.

ELIGIBILITY:
Inclusion Criteria:

* Children (0-18 years old) attending the paediatric ED or who are inpatients on the paediatric wards at STSFT

Exclusion Criteria:

* Critically ill children (judged so by treating physicians), including unconscious children
* Children who are non-compliant in terms of excessive movement during the measurement
* Children of parents/guardians/carers who are non-English speakers

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: We will be recruiting 500 child participants in the paediatric emergency department (PED) and hospital wards. The number will also include particiapnts for sub-protocols to measure blood pressure and record an electrocardiogram (ECG) in compliant and eligible participants and to conduct post-measurement questionnaires.
  A pilot project involving up to 10% (50) participants will run for 3 weeks in advance of the study with the aim of identifying the most efficient and effective way to deliver the study activities.
Sampling Method: Non-Probability Sample
Enrollment: 504 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Overall outcome measure | 6 months
  Train Lifelight algorithms across more extensive paediatric clinical ranges in 500 subjects
Heart rate | 6 months
  The following accuracy metrics are indicative minimum performance requirements for Lifelight® Junior. VISION-Junior should progress the technology towards these performance targets:
  • Heart rate
  o Root mean square error of 5 bpm or lower
Respiratory rate | 6 months
  The following accuracy metrics are indicative minimum performance requirements for Lifelight® Junior. VISION-Junior should progress the technology towards these performance targets:
  • Respiratory rate
  o Maximum error of 5 breaths per minute for 100% of the measurements
Oxygen saturation level (percentage) | 6 months
  The following accuracy metrics are indicative minimum performance requirements for Lifelight® Junior. VISION-Junior should progress the technology towards these performance targets:
  • Oxygen saturation
  o Maximum error tolerance of 4%.

CONTACTS AND LOCATIONS:
Overall Officials: Niall Mullen, MB BCh, Principal Investigator — South Tyneside and Sunderland Foundation Trust
Locations (1):
- South Tyneside and Sunderland NHS Foundation Trust, Sunderland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Misra G, Wegerif S, Fairlie L, Kapoor M, Fok J, Salt G, Halbert J, Maconochie I, Mullen N. The Measurement of Vital Signs in Pediatric Patients by Lifelight Software in Comparison to the Standard of Care: Protocol for the VISION-Junior Observational Study. JMIR Res Protoc. 2025 Mar 14;14:e58334. doi: 10.2196/58334. PMID 40085833